CLINICAL TRIAL: NCT00178295
Title: Radiation-Induced Cytokine Cascades and Their Correlation With Central Nervous System Injury
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Louis Constine, Principal Investigator, University of Rochester
Other Study IDs: URCC 11095
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Brain Neoplasm
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood plasma
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Radiation Therapy — standard of care for the cancer being treated

SUMMARY:
Treatment for brain cancer may include radiation therapy. Radiation therapy is the treatment of tumors with X-rays. This study is related to understanding the side effects of radiation treatment for brain tumors.

This study is being conducted by the University of Rochester Cancer Center to compare the extent of side effects of brain cancer treatment with changes in levels of blood proteins called cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who will be treated to the brain or spinal axis for a CNS tum Patients so treated will be stratified according to whether or not the hypo is included in the treatment fields.
* Patients receiving external beam radiation to the brain may also be rece chemotherapy or interferon-beta. (Add. #1, 11-9-95)
* Patients receiving high dose rate (stereotactic radiosurgery) are eligible.
* Patients must sign a study specific informed consent meeting all federal a guidelines.
* Patients of any age, including children, are eligible (Add. #3, 11/25/97).

Exclusion Criteria:

* Patients who have a malignancy involving the hypothalamic-pituitary ax
* Patients who are not treated with irradiation to the brain or spinal axis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient who are going to receive radiation therapy as part of the treatment for their brain cancer
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 1999-11; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Cytokine blood levels | 12 weeks from start of radiation

CONTACTS AND LOCATIONS:
Overall Officials: Louis S Constine, MD, Study Chair — Universtiy of Rochester, Dept of Radiation Oncology; Ralph Brasacchio, MD, Study Chair — University of Rochester, Department of Radiation Oncology
Locations (1):
- University of Rochester, Dept. Radiation Oncology, Rochester, New York, United States